CLINICAL TRIAL: NCT06023108
Title: A Single Center,Randomized,Controlled Trial Assessing the Effects of Spectacles or Orthokeratology on Dry Eye Parameters in Children and Adolescents.
Brief Title: Assess the Effects of Spectacles or Orthokeratology on Dry Eye Parameters in Children and Adolescents.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: orthokeratology 2023
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye Disease
Keywords: Myopia; Orthokeratology; Tear film; Dry eye
MeSH Terms: conditions — Dry Eye Syndromes; Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthokeratology group (Experimental): Participants in OK lenses group will wear OK lenses at least 8 hours per day for 12 months.
  Interventions: Device: Orthokeratology
- Spectacles group (Active Comparator): Participants in spectacles group will wear per day for 12 months.
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Orthokeratology — OK lenses will be used to evaluate the condition that causes dry eye in the treatment of myopia.
  Other Names: OK lenses
  Arms: Orthokeratology group
Device: Spectacles — Spectacles will be used to evaluate the condition that causes dry eye in the treatment of myopia.
  Arms: Spectacles group

SUMMARY:
Orthokeratology(OK) is currently one of the effective methods for treating myopia, reshaping the corneal epithelium to change refractive power. Due to its contact with the ocular surface, long-term wearing could lead to symptoms and signs of dry eye disease(DED) , as well as changes in tear film stability. This prospective study randomly divided 300 children and adolescents with myopia into OK group and spectacles group, with a follow-up of 12 months. At baseline, 1, 3, 6, and 12 months, non-invasive tear breakup time (NIBUT), ocular surface disease index (OSDI) and visual analogue score (VAS) score, tear meniscus height (TMH), conjunctival hyperemia (RS score) and meibomian gland (MG) scores, tear MMP-9 concentration, and point-of-care Lymphotoxin alpha (LTA) test.

DETAILED DESCRIPTION:
This study will be conducted in compliance with the tenets of the Declaration of Helsinki and the Institutional Review Board of He Eye Specialist Hospital, Shenyang, China [ethics approval number:

In recent years, the prevalence of myopia has significantly increased nationwide, The incidence rate of myopia among adolescents in China has risen significantly, causing blurred vision. Severe myopia can cause complications that threaten vision, such as glaucoma and macula disease. It would be highly undesirable to increase the social burden. Myopia can be corrected by orthokeratology (OK) and spectacles. It has been shown in numerous researches that orthokeratology lens are recognized as one of the effective methods in the treatment of myopia, has been widely used nationwide. In current years, the clinical treatment of myopia by OK lens in adolescents are increasingly confirmed to prevent the progression. Traditional OK lenses change refractive power by reshaping the corneal Epithelium (leading to the redistribution of corneal epithelium). As the overnight OK lens directly contact the ocular surface, the patients may endure symptoms and signs of dry eye disease (DED), which may even have some impact on the health of the ocular surface, including potential complications such as Keratitis. In addition, corneal staining often has occurred in ook wearers. According to previous studies, it has shown that wearing contact lens will affect the tear film stability, damage the function of the meibomian gland, tear film thinning, its affect ocular inflammation. Recent studies have also shown that OK continuous wearing has the least impact at 12 months. In order to ensure the safety of long-term wearing ok lenses in children and adolescents, the effect of OK lens on tear film and meibomian gland demonstrated further exploration.

The aim of this study is to evaluate the effect of OK on the ocular surface and meibomian gland function in children and adolescents. To assess the effect of OK on ocular surface and meibomian gland function in children and adolescents, so as to improve the application of the clinical.

ELIGIBILITY:
Inclusion Criteria:

(i)myopia up to -5.5D; and with-the-rule astigmatism of up to 1.5 DC or against-the rule astigmatism of <-0.5DC with keratometry from 40 to 45D ; (ii)participants and guardians agree to be randomly assigned and are willing to cooperate with doctors for follow-up and examination.

Exclusion Criteria:

(i) existing ocular trauma, infectious diseases, recent surgical history; (ii) keratitis or any ocular inflammation or infection; recently wearing contact lenses; allergy history; (iii) glaucoma, active uveitis or retinal disease; (iv) systemic diseases.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-11-23 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear break-up time | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
OSDI Score | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  Chinese translated, and validated OSDI (Allergan Inc, Irvine, USA) version will be used to assess and quantify DE symptom. The 12 items of the questionnaire can be tabulated into a score that ranges from 0 (no symptoms) to 100 (severe symptoms) points.
VAS score | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  VAS is used to evaluate subjective symptoms, such as patient symptoms, emotions, etc. Composed of a 100 mm straight line, the end is defined as the limit of pain to be measured, resulting in a 100 component scale. The patient rated their eye discomfort by marking the continuity from 'no eye discomfort' (score 0) to 'my eye discomfort is as bad as ever' (score 100).

SECONDARY OUTCOMES:
Tear meniscus height (TMH) | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  Tear meniscus height using the Keratograph 5M (Oculus, Germany) topographer
Conjunctival hyperemia (RS score) | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  Conjunctival hyperemia (RS score) will be assessed by keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 to 4.0.
Meibomian gland score (meiboscore) | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  Meibomian gland score will be assessed by keratograph image (Oculus, Germany) .The meibomian gland can be scored that ranges from grade 0 (no loss) to grade 3 (more than two third loss).
MMP-9 detection | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  Inflammation Dry, (Rapid Pathogen Screening Inc., Sarasota, FL, USA) is a patented and proprietary modification of a traditional lateral flow device and uses direct sampling microfiltration technology.
LTA | Day-0 (baseline), 1-month ,3-month,6-month and 12-month.
  LTA will be measured using an immunochromatography assay by collecting 1ul tear samples from the lateral canthus using a capillary tear collector. To assess the concentration of LTA in the tear samples, a commercial reagent card (S05B, Seinda Biomedical Corporation, Guangdong, China) based on colloidal gold and immunochromatographic analysis was utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric E Pazo, PHD, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
The study's findings will be shared regardless of the effect's direction. All possible beneficiaries of the research, including patients, carers, family, doctors, advisory boards, and medical boards, will receive trial data. Publications in high-impact, open-access medical journals and talks at national and international medical conferences will serve this purpose.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Tao Z, Wang J, Zhu M, Lin Z, Zhao J, Tang Y, Deng H. Does Orthokeratology Wearing Affect the Tear Quality of Children? Front Pediatr. 2022 Jan 18;9:773484. doi: 10.3389/fped.2021.773484. eCollection 2021. PMID 35118029
- [Result] Hui W, Xiao-Feng H, Song-Guo L, Jing-Jing W, Xuan H, Yong T. Application of orthokeratology on myopia control and its effect on ocular surface and meibomian gland function in Chinese myopic adolescents. Front Med (Lausanne). 2022 Dec 8;9:979334. doi: 10.3389/fmed.2022.979334. eCollection 2022. PMID 36569150
- [Result] Yan ZP. Dry eye symptoms and signs in children wearing OK lenses for six months in China. J Fr Ophtalmol. 2020 Mar;43(3):211-215. doi: 10.1016/j.jfo.2019.07.029. Epub 2020 Jan 27. PMID 32000988
- [Result] Fricke TR, Holden BA, Wilson DA, Schlenther G, Naidoo KS, Resnikoff S, Frick KD. Global cost of correcting vision impairment from uncorrected refractive error. Bull World Health Organ. 2012 Oct 1;90(10):728-38. doi: 10.2471/BLT.12.104034. Epub 2012 Jul 12. PMID 23109740
- [Result] Kakita T, Hiraoka T, Oshika T. Influence of overnight orthokeratology on axial elongation in childhood myopia. Invest Ophthalmol Vis Sci. 2011 Apr 6;52(5):2170-4. doi: 10.1167/iovs.10-5485. PMID 21212181
- [Result] He M, Du Y, Liu Q, Ren C, Liu J, Wang Q, Li L, Yu J. Effects of orthokeratology on the progression of low to moderate myopia in Chinese children. BMC Ophthalmol. 2016 Jul 27;16:126. doi: 10.1186/s12886-016-0302-5. PMID 27464993
- [Result] Nti AN, Berntsen DA. Optical changes and visual performance with orthokeratology. Clin Exp Optom. 2020 Jan;103(1):44-54. doi: 10.1111/cxo.12947. Epub 2019 Aug 4. PMID 31378996
- [Result] Wang X, Li J, Zhang R, Li N, Pang Y, Zhang Y, Wei R. The Influence of Overnight Orthokeratology on Ocular Surface and Meibomian Gland Dysfunction in Teenagers with Myopia. J Ophthalmol. 2019 Jan 21;2019:5142628. doi: 10.1155/2019/5142628. eCollection 2019. PMID 30805209
- [Result] Yang L, Zhang L, Jian Hu R, Yu PP, Jin X. The influence of overnight orthokeratology on ocular surface and dry eye-related cytokines IL-17A, IL-6, and PGE2 in children. Cont Lens Anterior Eye. 2021 Feb;44(1):81-88. doi: 10.1016/j.clae.2020.04.001. Epub 2020 Apr 30. PMID 32359968
- [Result] Yu H, Yuan Y, Wu W, Zeng W, Tong L, Zhang Y, Feng Y. Orthokeratology Lens Wear for 2 Years in Children Did Not Alter Tear Film Lipid Thickness by Non-Invasive Interferometry. Front Med (Lausanne). 2022 Feb 10;9:821106. doi: 10.3389/fmed.2022.821106. eCollection 2022. PMID 35223920
- [Result] Lee J, Hwang G, Ha M, Kim HS, Han K, Na KS. Evaluation of the meibomian glands using the tear interferometer wearing orthokeratology lenses. BMC Ophthalmol. 2022 Mar 24;22(1):133. doi: 10.1186/s12886-022-02365-3. PMID 35331178
- [Derived] Song Y, Chen J, Qin G, Xu L, He W, Yu S, Pazo EE, He X. A protocol for a single center, randomized, controlled trial assessing the effects of spectacles or orthokeratology on dry eye parameters in children and adolescents. Heliyon. 2024 Sep 12;10(18):e37779. doi: 10.1016/j.heliyon.2024.e37779. eCollection 2024 Sep 30. PMID 39323780